CLINICAL TRIAL: NCT06618417
Title: National Decentral/Virtual Randomized Trial Testing Remote Sleep Apnea Evaluation in Patients with Atrial Fibrillation
Brief Title: Evaluating the Impact of Home-Based Sleep Apnea Diagnostic on Well-Being, Health Behavior, and AF Load in Patients with Atrial Fibrillation Using a Decentralized Platform
Acronym: VIR-SAAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Morten Lamberts, Associate Professor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023-12410
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF); Sleep Apnea
Keywords: atrial fibrillation; decentralized; sleep apnea home-evaluation; randomized; digital health; quality of life
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention will be sleep apnea home-evaluation
  Interventions: Device: sleep apnea home-evaluation
- Control (No Intervention): This arm will not undergo sleep apnea home-evaluation

INTERVENTIONS:
Device: sleep apnea home-evaluation — Participants will receive a home-monitoring device by mail to test for sleep apnea at home
  Other Names: sleep apnea diagnostics
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to find out if testing for sleep apnea (a condition where breathing stops and starts during sleep) at home can improve well-being in people with atrial fibrillation (an irregular heartbeat condition). About 936 participants will be involved. They will either be tested for sleep apnea and treated, if needed, or not tested at all.

Researchers will compare the well-being and heart-related symptoms of participants who are tested for sleep apnea to those who are not. These will be tracked using a mobile app to monitor symptoms, physical activity, and heart rhythm.

Main hypothesis: Participants with atrial fibrillation who are tested and possibly treated for sleep apnea will have improved quality of life scores (measured by the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire) by at least 5 points after 18 weeks.

DETAILED DESCRIPTION:
Background &amp;amp;amp; Clinical Relevance Atrial fibrillation (AF) is often described as reaching epidemic proportions. On a societal level, methods using new technology are needed as hospitals and payers need to rethink how to manage future care for patients with AF. For the patient, risk factor management is crucial to ensure optimal care, lowering the burden of hospitalizations, promoting physical and mental health behavior and increasing Quality of Life (QoL).

In recent years an integrated approach to management of AF has been recommended including focus on optimal risk factor evaluation such as hypertension, diabetes, smoking, and obesity. Presence of obstructive SA in relation to AF has recently also been established as an important modifiable risk factor. SA refers to intermittent, cessations or reductions of airflow during sleep and is accompanied by hypoxia, sleep arousals, and hemodynamic changes. The most prevalent form is obstructive sleep apnea (SA) with partial or complete collapse of the upper airway. OSA activates the sympathetic nervous system during respiratory events. This potentiates vasoconstriction which often triggers an increase in blood pressure and heart rate which is the suggestive mechanism behind the link to AF. The diagnosis of SA is based on the number of apneas and hypopneas per hour of sleep, i.e. the Apnea-Hypopnea Index (AHI). SA is categorized as mild (5-14 AHI), moderate (15-29 AHI) or severe (≥ 30 AHI).

Some centers report up to 85% of AF patients having SA, and our 126-patient study of an all-comer Danish population shows 56% with moderate to severe SA, which should be eligible for treatment. SA treatment typically includes continuous positive airway pressure (CPAP) if moderate or severe SA is present (i.e. an AHI of &amp;amp;amp;amp;amp;amp;amp;gt;15 per hour). Interestingly, presence of SA has not been given the same attention as ensuring adequate blood pressure, weight control or diabetes management in AF. Despite this, overwhelming evidence suggests that AF patients with OSA receiving CPAP treatment are less likely to have AF recurrences after 12 months following cardioversion compared to AF patients not receiving CPAP treatment. Additionally, several nonrandomized observational studies indicate that CPAP can help maintain sinus rhythm after ablation in patients with AF who have OSA, and need for antiarrhythmic drugs are less needed in CPAP treated AF patients . Due to daytime sleepiness and fatigue, SA in itself may be a possible causal factor for physical inactivity and in addition lowering general state of health.

These findings highlight that SA is critically unrecognized and therefore undertreated, particularly in patients with AF. Current guidelines recommend screening of AF (IIa recommendation) in patients with SA, but unclear on how to approach SA in AF patients in terms of how and when to test for SA. Though SA is a trigger for cardiac arrhythmia and a substrate for AF maintenance and progression, it is uncertain if systematic screening of SA in patients with AF is beneficial. Importantly, it has been shown that standard SA screening questionnaires fail to capture high-risk individuals with AF and consequently the benefit in a larger scale SA evaluation is poor. The gold standard of SA diagnosis with polysomnography (PSG) or cardiorespiratory monitoring (CRM) is information rich but is cumbersome, time-consuming and not widely available. Several sensors and belts measuring posture, chest movement, abdominal movement and nasal airflow are used. Often it includes an overnight stay or at least three hospital visits (instruction for application, return of the device and follow-up visit for the results).

Therefore, a new approach to manage AF patients for SA evaluation including estimating the clinical effect is needed. A proof-of-concept of a virtual management pathway has recently been suggested which are incorporated in this proposal. In VIRTUAL-SAFARI, AF patients awaiting ablation were offered education on the impact of concomitant OSA followed by information on a virtual sleep-disordered breathing project setup. The setup included digital referral to virtual sleep laboratory, home sleep test, results and data submission, virtual consultation, and CPAP treatment in the majority of the app. 50% diagnosed with SA. Indeed, emerging new technologies consisting of miniaturized monitoring devices and accurate algorithm development may transform how patients and clinicians approach risk factor management. Together with increased awareness from regulators of the benefits of virtual (or decentralized) trials (i.e. reduced or no site visits from patients) in the COVID era, current research practice but also future patient management need to consider how incorporating innovative methods can improve care, patients-related outcomes and prognosis. Notably, it is paramount when implementing new patient care pathways that evidence is based on unbiased and independent research and not pushed by commercial or industrial stakeholders. Our pilot trial, Mini VIR-SAAF, successfully demonstrated the feasibility of a completely decentralized clinical trial setup, confirming the proof of concept with the inclusion of 20 participants. The use of home-evaluation for SA, physical tracking and heart rhythm monitoring was well-received, with only one participant dropping out. This low drop-out rate indicates strong participant engagement and satisfaction. Given these positive results, the investigators are confident in scaling up the project to a national level, building on the insights gained to further optimize participant onboarding and study commitment.

Study Design This is an investigator-initiated virtual (or decentralized) trial that includes a postal parcel (mail-in) containing sensors for SA diagnosis (WatchPAT One) and physical activity (SENS Motion), in addition to smart-phone based heart rhythm (FibriCheck) monitoring in participants with paroxysmal or persistent AF. A case-coordinator (the investigators) will manage all participant contacts virtually during the study from inclusion to follow-up.

Sign-up for inclusion Participants interested in participating in the study can sign up on our website, www.vir-saaf.dk. In the registration form, participants will be asked to provide their full name, email, phone number, and the region they live in. Additionally, they will be asked if they have been diagnosed with AF and if they have ever undergone any SA testing. This information will serve as an initial screening for study eligibility. The data collected from the registration form will be securely stored in RedCap.

Inclusion:

After signing up on the webpage, participants will be called by telephone by the investigators to be further informed of the study. Subsequently, participants will be invited to the Introduction Video Meeting via an SMS with a link to a video meeting. At the Introduction Video Meeting, the participants will receive oral information about the study. Also digital written information with full details of the study ("Deltager information" and "Før du beslutter dig"), including risks and benefits, will be available to potential participants. Please see the section "Recruiting and Giving Consent" below for a detailed description of obtaining informed consent from participants.

After the Introduction Video Meeting, eligible participants accepting to participate will be able to download our application, through which written informed consent via MitID will be obtained. Once consent has been given, final confirmation of study eligibility will be performed by entering key variables into a secure web-based program (RedCap) at the Cardiovascular Research Center at Herlev-Gentofte Hospital.

After inclusion, participants who answer digital questionnaires (Survey 1) will receive a mail-in package containing either the WatchPAT One device and the SENS Motion device (intervention group) or only the SENS Motion device (control group). The Survey 1 will include basic participant information (such as email, address, height, weight, self-measured neck circumference [important measurement in sleep apnea], and employment status [important factor to assess physical activity patterns]) and the following questionnaires: Atrial Fibrillation Effect on QualiTy-of-life (AFEQT), AF Severity Scale (AFSS), Pittsburgh Sleep Quality Index (PSQI), and The eHealth Literacy Questionnaire (eHLQ). Please see document 08.01 for the complete questionnaires.

Furthermore, a clinical evaluation form will be filled out by the investigators based on electronic charts or from the Introduction Video Meeting, which includes: CPR number, sex, birth date, questions related to AF (modified European Heart Rhythm Association (mEHRA) symptom classification (0-4)), concomitant CVD medication (antithrombotic medication, rate-lowering drugs, anti-arrhythmic drugs), date of first AF detected, type of AF (paroxysmal or persistent AF), and other relevant medical conditions.

Randomization Automatic patient randomization in the two arms (ratio 2:1) will be performed in R-studio. The randomization key will be stored in a locked and secure environment at the Cardiovascular Research Center at Gentofte Hospital. The primary endpoint will be evaluated and determined by an independent committee blinded to randomization.

Postal Parcel 1:

After completing Survey 1, a postal parcel (postal parcel 1) including either the WatchPAT One device and the SENS Motion (intervention) or only the SENS Motion (control) will be sent to the participant's address. The postal parcel 1 will also include detailed written information and instructions for the devices and applications together with a user-friendly written overview of the study design. As soon as the participants receive the postal parcel 1, the participant will begin their home monitoring with the 1 night of WatchPAT One monitoring (only intervention group), the 7 days of activity tracker (round 1) with SENS Motion, and daily heart rhythm monitoring with the FibriCheck application.

During the home monitoring, if the participants have any questions, concerns or difficulties using devices or applications, a telephone number will be given to contact the investigators directly. Also, a frequently-asked question section is made available to the participants in the VIR-SAAF trial app.

Return of equipment 1:

After completing the 7 days of activity tracker round 1 with SENS Motion, the participants will ship the used SENS Motion device back to the investigators. This will be done via a prepaid shipping label for Department of Cardiology, Copenhagen University Hospital Herlev and Gentofte, Gentofte Hospitalsvej 1, 2900 Hellerup. The WatchPAT One is a disposable (intervention group) and the participants receiving the device are thoroughly informed how to discard the device correctly (electronic waste). No data is stored on the device.

SA evaluation in cooperation with the Danish Center for Sleep Medicine, Glostrup:

Participants in the active arm will be scheduled for a SA Evaluation Video Meeting with the investigators.

In case the evaluation shows no or only mild SA the participants are informed that the evaluation did not show any signs of significant SA. If a participant reports a major degree of symptoms that could be a result of SA, a referral to a sleep physician will be done.

In case the evaluation shows moderate to severe SA, the participants are informed that the evaluation shows signs of significant SA that should be evaluated for indication for treatment. If accepting, the participants will be referred to a sleep physician for clinical assessment of diagnosis and potential treatment.

Dansk Center for Søvnsygdomme (Glostrup Hospital, Copenhagen) will be the primary center for the clinical assessment. However, local sleep centers, if accepted, will also be involved in the clinical assessment and responsible for initiating CPAP treatment (based on clinical assessment and judgment).

Postal Parcel 2:

At week 15, a postal parcel (postal parcel 2) with the SENS Motion will be sent to the participants' address for activity tracking (round 2). As soon as the participants receive the postal parcel 2, the participant will begin their 7 days of activity tracker round 2 with SENS Motion.

Return of equipment 2:

After completing the 7 days of activity tracker round 2 with SENS Motion, the participants will ship their used device back to the investigators. This will be done via a prepaid shipping label.

Follow up:

After completing the 7 days of activity tracker round 2, questionnaires (Survey 2) will once again be pushed digitally to participants including AFEQT, AFSS, PSQI and eHLQ.

At week 19 the participant will be scheduled for an End of Study Video Meeting where the participant's own study results will be presented.

During follow-up, if the participants have any questions, concerns or difficulties using devices, a telephone number will be given to contact the investigators directly.

Post-study Follow up:

After the conclusion of the study, participants will receive a long-term follow-up survey 9 months later, which will include the same questionnaires previously administered. These will be sent via email or Digital Post. This follow-up is not an extension of the study but rather a separate effort to gather valuable data on the sustained effects of the interventions.

Devices and Questionnaires SA evaluation by WatchPAT One Only participants in the intervention group will by postal parcel 1 receive a SA evaluation device (WatchPAT One) to be evaluated for SA by 1 night of recording after completing the Survey 1.

The WatchPAT One system can via a validated algorithm derive all diagnostic parameters recommended by The AASM Manual for the Scoring of Sleep and Associated Events for home SA testing. It has been validated against polysomnography with a very close agreement when estimating AHI.

Physical activity tracking by SENS Motion All participants will after completion of Survey 1 be receiving a SENS Motion device for tracking physical activity through postal parcel 1. The tri-axial accelerometer is to be worn laterally on the thigh in 7 days. The participants will be using the accelerometer for 7 days. The device can store up to 10 days of physical activity data.

At week 18, all participants will be receiving postal parcel 2 with a new SENS Motion device for activity tracker round 2. The postal parcel 2 will only be containing the SENS Motion device.

Heart rhythm monitoring by FibriCheck application All participants will after completion of Survey 1 start using the FibriCheck application for evaluating AF recurrence by monitoring heart rhythm two times a day (morning and evening) and in the case of symptoms throughout the study period. The solution is based on a validated algorithm following participants holding their index finger on their smartphone camera for one minute.

Digital questionnaires All participants will be filling out questionnaires digitally through RedCap. This includes AFEQT. The score ranges from 0 (worst) to 100 (best) based on 20 questions on a seven point Likert Scale. The AFEQT covers AF symptoms, daily activities and treatment concerns within the last 4 weeks. AFEQT has been validated in various settings. Also AFSS will be evaluated. AFSS is more focused on AF symptoms and captures subjective and objective ratings of AF related symptoms, health care utilization, and AF disease burden. Sleep will be measured by PSQI. These three questionnaires will also be filled out at the end of the study period (after 3 months) for estimating the effect of the SA evaluation. Furthermore, the same three questionnaires will be pushed once again a month after the end of the study period.

At the start of the study all participants will also be asked to fill out the eHealth Literacy Questionnaire (eHLQ). This model consists of 7 dimensions, which describes the attributes of the users (information and knowledge about their health); the intersection between users and the technologies (their feeling of being safe and in control and their motivation); and users experience of systems (they work and are accessible, and suits users' needs). The method will give us a more nuanced picture of participants´s digital health literacy prior to participating in a virtual trial.

Statistical analysis of data Sample size and primary endpoint The investigators will assess 2:1 randomization of mail-in WatchPat One home-evaluation versus no home evaluation. The randomization ratio is selected to provide a larger "treatment" group for further evaluation and to ensure improved recruitment. The final sample size will be calculated based on a clinically relevant 5-point difference in AFEQT score (margin) at 18 weeks (primary endpoint). Estimated target of 936 patients (624 active arm, 312 in control arm) with a power of 80% and assumed standard difference (SD) of 22 based on the pilot study. A maximal drop-out rate of 10% is included

Analysis of data The investigators will include data from all participants in the analyses of the primary and secondary endpoints according to the intention-to-treat principle. Baseline characteristics are summarized as means and standard deviations, medians and interquartile ranges, or percentages. Primary endpoint of AFEQT score will be evaluated by assessing mean outcome values between the intervention and control group at baseline and 18 weeks by repeated measures analysis of variance (ANOVA). Point estimates for each intervention group and mean estimates difference with 95% CI will be calculated at 18 weeks. The secondary endpoint of AF load at 18 weeks will be measured after 6 weeks from inclusion, and percentage of measurements with PPG-documented AF of all measurements performed from week 7 to week 18 will be calculated. Any missing data will be replaced by a proximate examination from a prespecified imputation algorithm. The secondary endpoint for physical activity tracking will be comparison of time spent physical inactivity between control and intervention group. The difference in physical inactivity will be tested using repeated measures ANOVA. A predefined stratification between work and leisure time will be included in the analysis. A significance level of 0.05 will be used.

Recruiting and giving consent All potential participants will be contacted by investigators after signing up on the website www.vir-saaf.dk by a phone call. In the phone call the participants will receive a short introduction to the study and screening for eligibility. During the phone call the participant will also agree on a time for the Introduction Video Meeting. After the call, the participants will receive a SMS with an invitation link to the scheduled Introduction Video Meeting. The Introduction Video Meeting will be held with the VDX application or other approved solution. Digital written information with full details of the study, including risks and benefits, will be available for the participants before the scheduled Introduction Video Meeting on the website www.vir-saaf.dk. Participants will also be informed of their right to have an assessor present at the Introduction Video Meeting. Prior to the Introduction Video Meeting, a video about the purpose of the study, study design, participant requirements, and the devices used will be made available to participants. This will ensure that participants can prepare questions beforehand and identify any aspects of the study design that require further clarification. Eligible patients with AF will receive verbal information about the study during the Introduction Video Meeting. The oral and written information will include details regarding the postal parcels participants will receive, as well as comprehensive information on the devices and questionnaires used in the study. The investigators require written consent from all eligible participants prior to their inclusion in the study. Only the investigators will be allowed to obtain informed consent and provide oral information about the study. Before signing the informed consent form, the investigator will ensure during the Introduction Video Meeting that the participant has read and understood the written and verbal study information.

All participants will be offered up to 24 hours to consider their options, having a friend or family member present, and the participants will be given every opportunity to reverse their decision to enroll in the study.

The written informed consent gives the control authority direct access to the participant's journal, including electronic chart, for the purpose of acquiring information about the participant's health condition that allows for quality control, control of adherence to study protocol and monitoring of the study (all which is mandatory for clinical research projects). Researchers affiliated to the project obtain necessary information in the participant's journal, such as medication, prior health conditions (comorbidities), prior examinations performed, and blood tests. The researchers will only use access to the electronical participants charts until any subsequent work-up for SA has finished or 12 months following inclusion. All patient related information will be directly transferred to the specific project RedCap database.

Ethics The trial is conducted in accordance with ethical principles of the Declaration of Helsinki. Management and documentation of data will be handled according to Guidelines for Good Clinical Practice. Appropriate local regulatory approvals have been granted. Personal sensitive data will be handled according to local and national requirements. Following study completion, the database will be closed for statistical analyses, interpretation and submission to scientific journals. Furthermore, the database will be anonymized and transferred to closed servers at Statistics Denmark for further research.

WatchPAT, FibriCheck and SENS Motion are CE marked and comply with general requirements and technical standards for medical devices (IEC 60601-1).

ELIGIBILITY:
Inclusion Criteria:

* Established paroxysmal or persistent AF diagnosis
* Owning a compatible smartphone (or accepting a smart phone provided by the investigators)
* Understanding of potential SA treatment possibilities including CPAP treatment

Exclusion Criteria:

* Previous investigation for sleep-disturbed breathing
* Advanced heart failure (left ventricular dysfunction and NYHA III/IV)
* Occupational driver licenses
* Pregnancy
* Doxazosin or Terazosin (alpha-adrenergic antagonists)
* Peripheral arterial disease with daily intermittent claudication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 18 weeks
  The primary outcome is the Atrial Fibrillation Effect on Quality-Of-Life (AFEQT) questionnaire, which scores from 0 (worst) to 100 (best), based on 20 questions using a seven-point Likert scale.

SECONDARY OUTCOMES:
AF load | 18 weeks
  AF load by heart rhythm measurement using Fibricheck. The solution is based on a validated algorithm following patients holding their index finger on their smartphone camera during one minute. Participants will be asked for heart rhythm measurements morning, evening and in case of AF symptoms.
Physical health behavior | 18 weeks
  Physical activity will be measured by a tri-axial accelerometer (SENS Motion) worn at the lateral of the thigh for 7 days. From the accelerometer data time spent physical inactive (minutes/day) will be calculated
Symptom severity | 18 weeks
  AF severity scale (AFSS) questionnaire. AFSS is focused on AF symptoms and captures subjective and objective ratings of AF related symptoms, health care utilization, and AF disease burden. The questionnaire scores from 0 (best) to 35 (worst).

OTHER OUTCOMES:
Hospitalization and ablation | 5 years
  Long-term AF hospitalization and ablation following linkage with health registers.
Sleep quality | 18 weeks
  Pittsburgh Sleep Quality Index (PSQI) to distinguish good and poor sleepers. The questionnaire's global score range from 0 (best) to 21 (worst).
Quality of Life - Long-term follow up | One year
  One year after randomization, participants will complete the Atrial Fibrillation Effect On Quality-Of-Life (AFEQT) questionnaire again to assess the long-term effects of home-based sleep apnea evaluation. The score ranges from 0 (worst) to 100 (best).
Digital Health literacy | 18 weeks
  The eHealth Literacy Questionnaire (eHLQ) to assess digital health literacy before and after the study to measure potential changes. Scores is calculated as a mean from the 7 different dimensions in the questionnaire. The score ranges from 1 to 4 with higher values indicating better eHealth literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fein AS, Shvilkin A, Shah D, Haffajee CI, Das S, Kumar K, Kramer DB, Zimetbaum PJ, Buxton AE, Josephson ME, Anter E. Treatment of obstructive sleep apnea reduces the risk of atrial fibrillation recurrence after catheter ablation. J Am Coll Cardiol. 2013 Jul 23;62(4):300-5. doi: 10.1016/j.jacc.2013.03.052. Epub 2013 Apr 23. PMID 23623910
- [Background] Linz D, McEvoy RD, Cowie MR, Somers VK, Nattel S, Levy P, Kalman JM, Sanders P. Associations of Obstructive Sleep Apnea With Atrial Fibrillation and Continuous Positive Airway Pressure Treatment: A Review. JAMA Cardiol. 2018 Jun 1;3(6):532-540. doi: 10.1001/jamacardio.2018.0095. PMID 29541763
- [Background] Mehra R, Chung MK, Olshansky B, Dobrev D, Jackson CL, Kundel V, Linz D, Redeker NS, Redline S, Sanders P, Somers VK; American Heart Association Electrocardiography and Arrhythmias Committee of the Council on Clinical Cardiology; and Stroke Council. Sleep-Disordered Breathing and Cardiac Arrhythmias in Adults: Mechanistic Insights and Clinical Implications: A Scientific Statement From the American Heart Association. Circulation. 2022 Aug 30;146(9):e119-e136. doi: 10.1161/CIR.0000000000001082. Epub 2022 Aug 1. PMID 35912643
- [Background] Verhaert DVM, Betz K, Gawalko M, Hermans ANL, Pluymaekers NAHA, van der Velden RMJ, Philippens S, Vorstermans B, Simons SO, den Uijl DW, Chaldoupi SM, Luermans JGLM, Westra SW, Lankveld T, Kadhim K, Pepin JL, van Steenwijk RP, Hol B, Schotten U, Sanders P, Vernooy K, Hendriks JM, Linz D. A VIRTUAL Sleep Apnoea management pathway For the work-up of Atrial fibrillation patients in a digital Remote Infrastructure: VIRTUAL-SAFARI. Europace. 2022 Apr 5;24(4):565-575. doi: 10.1093/europace/euab229. PMID 34718525
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Neilan TG, Farhad H, Dodson JA, Shah RV, Abbasi SA, Bakker JP, Michaud GF, van der Geest R, Blankstein R, Steigner M, John RM, Jerosch-Herold M, Malhotra A, Kwong RY. Effect of sleep apnea and continuous positive airway pressure on cardiac structure and recurrence of atrial fibrillation. J Am Heart Assoc. 2013 Nov 25;2(6):e000421. doi: 10.1161/JAHA.113.000421. PMID 24275628
- [Background] Patel D, Mohanty P, Di Biase L, Shaheen M, Lewis WR, Quan K, Cummings JE, Wang P, Al-Ahmad A, Venkatraman P, Nashawati E, Lakkireddy D, Schweikert R, Horton R, Sanchez J, Gallinghouse J, Hao S, Beheiry S, Cardinal DS, Zagrodzky J, Canby R, Bailey S, Burkhardt JD, Natale A. Safety and efficacy of pulmonary vein antral isolation in patients with obstructive sleep apnea: the impact of continuous positive airway pressure. Circ Arrhythm Electrophysiol. 2010 Oct;3(5):445-51. doi: 10.1161/CIRCEP.109.858381. Epub 2010 Aug 5. PMID 20689107
- [Background] Kanagala R, Murali NS, Friedman PA, Ammash NM, Gersh BJ, Ballman KV, Shamsuzzaman AS, Somers VK. Obstructive sleep apnea and the recurrence of atrial fibrillation. Circulation. 2003 May 27;107(20):2589-94. doi: 10.1161/01.CIR.0000068337.25994.21. Epub 2003 May 12. PMID 12743002
- [Background] Abumuamar AM, Dorian P, Newman D, Shapiro CM. The prevalence of obstructive sleep apnea in patients with atrial fibrillation. Clin Cardiol. 2018 May;41(5):601-607. doi: 10.1002/clc.22933. Epub 2018 May 10. PMID 29745973
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Corrigendum to: 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association of Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2021 Feb 1;42(5):507. doi: 10.1093/eurheartj/ehaa798. No abstract available. PMID 33029625
- [Background] Jons C, Hansen PS, Johannessen A, Hindricks G, Raatikainen P, Kongstad O, Walfridsson H, Pehrson S, Almroth H, Hartikainen J, Petersen AK, Mortensen LS, Nielsen JC; MANTRA-PAF Investigators. The Medical ANtiarrhythmic Treatment or Radiofrequency Ablation in Paroxysmal Atrial Fibrillation (MANTRA-PAF) trial: clinical rationale, study design, and implementation. Europace. 2009 Jul;11(7):917-23. doi: 10.1093/europace/eup122. Epub 2009 May 15. PMID 19447807
- [Background] Kayser L, Karnoe A, Furstrand D, Batterham R, Christensen KB, Elsworth G, Osborne RH. A Multidimensional Tool Based on the eHealth Literacy Framework: Development and Initial Validity Testing of the eHealth Literacy Questionnaire (eHLQ). J Med Internet Res. 2018 Feb 12;20(2):e36. doi: 10.2196/jmir.8371. PMID 29434011
- [Background] Lip GYH. The ABC pathway: an integrated approach to improve AF management. Nat Rev Cardiol. 2017 Nov;14(11):627-628. doi: 10.1038/nrcardio.2017.153. Epub 2017 Sep 29. No abstract available. PMID 28960189
- [Background] Isabelle C Van Gelder, Michiel Rienstra, Karina V Bunting, Ruben Casado-Arroyo, Valeria Caso, Harry J G M Crijns, Tom J R De Potter, Jeremy Dwight, Luigina Guasti, Thorsten Hanke, Tiny Jaarsma, Maddalena Lettino, Maja-Lisa Løchen, R Thomas Lumbers, Bart Maesen, Inge Mølgaard, Giuseppe M C Rosano, Prashanthan Sanders, Renate B Schnabel, Piotr Suwalski, Emma Svennberg, Juan Tamargo, Otilia Tica, Vassil Traykov, Stylianos Tzeis, Dipak Kotecha, ESC Scientific Document Group , 2024 ESC Guidelines for the management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): Developed by the task force for the management of atrial fibrillation of the European Society of Cardiology (ESC), with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Endorsed by the European Stroke Organisation (ESO), European Heart Journal, 2024;, ehae176, https://doi.org/10.1093/eurheartj/ehae176
- See also: Danish Health Authority — https://laegemiddelstyrelsen.dk/en/news/2021/guidance-on-the-implementation-of-decentralised-elements-in-clinical-trials-with-medicinal-products-is-now-available/~/media/5A96356760ED408CBFA9F85784543B53.ashx